CLINICAL TRIAL: NCT00575952
Title: A Phase I Study of IV Doxorubicin Plus Intraperitoneal (IP) Paclitaxel and IV or IP Cisplatin in Endometrial Cancer Patients at High Risk for Peritoneal Failure
Brief Title: Intraperitoneal Paclitaxel, Doxorubicin Hydrochloride, and Cisplatin in Treating Patients With Stage III-IV Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9920; NCI-2009-00623 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-9920; CDR0000580419; GOG-9920 (Other: NRG Oncology); GOG-9920 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Squamous Cell Carcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Carcinoma; Stage IIIA Uterine Corpus Cancer; Stage IIIC Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: interventions — Cisplatin; Doxorubicin; Filgrastim; Paclitaxel; pegfilgrastim

ARMS (1):
- Treatment (doxorubicin hydrochloride, cisplatin, paclitaxel) (Experimental): Patients receive doxorubicin hydrochloride IV over 30 minutes followed by cisplatin IV over 1 hour on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim SC on days 3-12 or pegfilgrastim SC on day 3. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients then receive doxorubicin hydrochloride IV and cisplatin IV or IP on day 1, and paclitaxel IP on days 1 or 8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Drug: Paclitaxel; Biological: Pegfilgrastim

INTERVENTIONS:
Drug: Cisplatin — Given IV or IP
Drug: Doxorubicin Hydrochloride — Given IV
Biological: Filgrastim — Given SC
Drug: Paclitaxel — Given IV or IP
Biological: Pegfilgrastim — Given SC

SUMMARY:
This phase I trial studies the side effects and best dose of intraperitoneal paclitaxel when given together with doxorubicin hydrochloride and cisplatin in treating patients with stage III-IV endometrial cancer. Drugs used in chemotherapy, such as paclitaxel, doxorubicin hydrochloride, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them in different ways may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of intraperitoneal (IP) paclitaxel when given concurrently with fixed dose intravenous (IV) doxorubicin (doxorubicin hydrochloride) and IV cisplatin.

II. To determine the maximum tolerated dose of IP paclitaxel when given concurrently with fixed dose IV doxorubicin hydrochloride and IP cisplatin.

III. To determine the feasibility of an IV/IP based doxorubicin hydrochloride, paclitaxel, and cisplatin chemotherapy regimen in patients with advanced endometrial cancer.

OUTLINE: This is a dose-escalation study of paclitaxel.

Patients receive doxorubicin hydrochloride IV over 30 minutes followed by cisplatin IV over 1 hour on day 1, paclitaxel IV over 3 hours on day 2, and filgrastim subcutaneously (SC) on days 3-12 or pegfilgrastim SC on day 3. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive doxorubicin hydrochloride IV and cisplatin IV or IP on day 1, and paclitaxel IP on days 1 or 8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IIIA, or stage IIIC with positive cytologic washings/ascites, adnexal spread, or serosal involvement, or stage IV (by virtue of intraperitoneal disease spread) histologically confirmed endometrial cancer (endometrioid, serous, clear cell, squamous/adenosquamous, undifferentiated, or mixed histologies)
* Patients must be optimally cytoreduced with less than or equal to 2 cm residual disease
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, equivalent to Common Toxicity Criteria (Common Terminology Criteria for Adverse Events [CTCAE] version 3.0 [v3.0]) grade 1
* Platelets greater than or equal to 100,000/mm^3 (CTCAE v3.0 grade 0-1)
* Hemoglobin greater than or equal to 10 g/dl (CTCAE v3.0 grade 1)
* Creatinine less than or equal to 2 mg/% or 24 hour creatinine clearance > 50 ml/min
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (CTCAE v3.0 grade 1)
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 x ULN (CTCAE v3.0 grade 1)
* Neuropathy (sensory and motor) less than or equal to CTCAE v3.0 grade 1
* Patients must have normal ejection fraction
* Patients must be enrolled within 8 weeks of surgery
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Metastatic disease involving lung or liver parenchyma, bone or inguinal or scalene lymph nodes
* Patients with GOG performance grade of 3 or 4
* Patients with concomitant medical illness such as serious uncontrolled infection, uncontrolled angina, or serious peripheral neuropathy, which in the opinion of the treating physician, makes the protocol prescribed treatments hazardous to the patient
* Patients with 3rd degree or complete heart block are not eligible unless a pacemaker is in place; patients who are on medications which alter cardiac conduction (digitalis, beta blockers, calcium channel blockers) or who have other cardiac conduction abnormalities may be placed on study at the discretion of the investigator
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiation or chemotherapy for the cancer being treated in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01-17 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

PRIMARY OUTCOMES:
Incidence of observed DLTs, defined as grade 3-4 hematologic or non-hematologic toxicity graded using CTCAE v3.0 | 18 weeks
Maximum tolerated dose (MTD) of IP paclitaxel with fixed dose IV doxorubicin hydrochloride and IV cisplatin, determined according to dose-limiting toxicities (DLTs) graded using CTCAE v3.0 | 12 weeks
MTD of IP paclitaxel with fixed dose IV doxorubicin hydrochloride and IP cisplatin, determined according to DLTs graded using CTCAE v3.0 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: D. McMeekin, Principal Investigator — NRG Oncology
Locations (9):
- United States (9):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island